CLINICAL TRIAL: NCT03459456
Title: Measuring Automated Behavioral Observations & Vocal Expressions (ABOVE) While Recording From the Brain
Brief Title: Measuring Automated Behavioral Observations & Vocal Expressions (ABOVE)
Acronym: ABOVE
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Brown University (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Wayne Goodman MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H41632
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: OCD; Obsessive-Compulsive Disorder
Keywords: OCD; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OCD subjects: Subjects meeting inclusion/exclusion criteria with OCD will be exposed to the following:
  * Provocation OC task (Provoc)
  * Trier Social Stress Test (TSST)
  * Exposure provocation task
  Interventions: Behavioral: Provocation OC task (Provoc); Behavioral: Trier Social Stress Test (TSST); Behavioral: Exposure provocation task
- Control subjects: Subjects meeting inclusion/exclusion criteria without OCD (age and gender matched with OCD subjects) will be exposed to the following:
  * Provocation OC task (Provoc)
  * Trier Social Stress Test (TSST)
  * Exposure provocation task
  Interventions: Behavioral: Provocation OC task (Provoc); Behavioral: Trier Social Stress Test (TSST); Behavioral: Exposure provocation task

INTERVENTIONS:
Behavioral: Provocation OC task (Provoc) — used to evoke OC-related distress
Behavioral: Trier Social Stress Test (TSST) — used to evoke anxiety unrelated to OCD (e.g., performance anxiety)
Behavioral: Exposure provocation task — used to elicit overt OCD rituals

SUMMARY:
The investigators propose to synchronize automated measurements of behavior - head, body, and face dynamics, gaze, and vocal prosody - with simultaneous recordings of brain activity in clinically relevant contexts.

DETAILED DESCRIPTION:
Baylor College of Medicine (BCM), University of Pittsburgh (UPitt) and Brown University will collaborate on this research project. BCM will be the only site that will enroll study subjects and perform study assessments. UPitt and Brown will supervise data management, measurement and modeling of multimodal signals and collaborate on research design and machine learning.

Following initial screening, subjects will participate in one testing session lasting about 2 hours. The addition of these preliminary studies will allow investigators to obtain information in order to differentiate and code OCD-distress versus social anxiety and identify rituals related to OCD.

Research Material, Data, and Information to be collected:

Interviews, rating scales, video, audio, behavioral assessments, and heart rate will be obtained.

Preliminary Testing in Un-implanted Subjects: Automated Behavioral Measures of OCD-related Distress (i.e., obsessions and urge to ritualize) and Overt Rituals:

The Provocation OC task (Provoc) and the Trier Social Stress Test (TSST) will be used to evoke OC-related distress and anxiety unrelated to OCD (e.g., performance anxiety), respectively. These tasks will be preceded by a neutral baseline (the subject may be asked to describe how they traveled to the clinic to the experimenter) and a positive affect induction, the Broad-Minded Affective Coping procedure (BMAC) a clinical technique that uses recalled positive autobiographical memories and mental imagery to elicit positive affect. Because anxiety and negative affect may have carryover effects, neutral baseline and BMAC will be presented prior to the non-OCD and OCD distress inductions. In the BMAC, subjects will be instructed to recall and describe a recent positive memory/experience. The order of Provoc and TSST will be counterbalanced across the subjects. Use of a conveyor belt may be used during the Provoc tasks to present the evoking stimuli. Simultaneously recorded measures are noted in the Table attached in Section S and include: AFAR, new suite of behavioral measures (shown as shaded), hand/arm movements and heart rate.

A third provocation task will be added to elicit overt rituals (e.g., handwashing) in the clinic. It will occur following the BMAC and TSST/Provoc tasks and a relaxation break.

Subjects will be asked to wash their hands at a sink in our clinic inside an exam room where their behaviors will be recorded using hardware-synchronized cameras: one, to capture frontal view of the face for AFAR; and another, to record full body movement for CPM. The investigators are aware of only one prior study of automated coding of compulsive behavior. In that study, a computer vision approach was able to discriminate subjects with OCD from healthy subjects on the basis of handwashing videos in which regions of interest (ROIs) were defined for objects (e.g., soap dispenser) used for handwashing. The investigators will combine this ROI paradigm with a CPM approach that captures hand and body movements. Dropouts from the ritual paradigm will be replaced.

These same tasks will also be performed on up to 4 subjects that have consented to receive a DBS implant on a separate protocol. Informed consent will also be collected from these implanted subjects for the purpose of completing the tasks described above on this study.

ELIGIBILITY:
Inclusion Criteria:

OCD subjects:

* The subject has a minimum score of ≥16 on the Y-BOCS;
* If applicable, on a stable pharmacologic regimen;
* Sample will be enriched with OCD subjects having contamination obsessions and handwashing compulsions, and scores on items 9 and 10 of the Y-BOCS reflecting difficulty resisting and controlling compulsions;

Healthy Control Subjects:

* Men and women will be age/gender matched with subjects
* Absence of any psychiatric disorder determined by the MINI^53 for DSM-5 with the exception of non-impairing specific phobia.
* Low scores on measures of contamination concerns and disgust sensitivity based on Y-BOCS scores below 10 and the Disgust Scale-Revised (total score <8).

Exclusion Criteria:

OCD Subjects:

* Subject has a documented lifetime diagnosis of psychotic disorders such as schizophrenia;
* Alcohol or substance abuse/dependence reported within 6 months, excluding nicotine;
* The subject is deemed at high risk of suicidal behavior or impulsivity. The Beck Depression Inventory^52 (BDI) will be completed by all subjects and responses reviewed by a clinician.

Healthy Control Subjects:

- Those not meeting the inclusion criteria described in the inclusion section above.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The primary source of OCD subjects will be self-referrals generated through BCM Clinicaltrials website, Clinicaltrials.gov, and BCM Psychiatry Clinic. The investigators also anticipate referrals from local area clinicians in addition to affiliate entities.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity | baseline to Hour 2
  measured before, during and after PROVOC task, Trier Social Stress Test (TSST) and exposure task

SECONDARY OUTCOMES:
Change in Heart Rate | baseline to Hour 2
  measured before, during and after PROVOC task, Trier Social Stress Test (TSST) and exposure task

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Goodman, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided